CLINICAL TRIAL: NCT03855969
Title: Frequency of Central Venous Port Catheter Removal Due to Suspected Infection in Patients Diagnosed With Cancer at a Single Institution: A Retrospective Study.
Brief Title: Central Venous Access Device Removal in Cancer Patients
Status: Completed | Type: Observational
Sponsor: General Hospital Groeninge (Other)
Responsible Party: Principal Investigator, Koen Van Eygen, Principle Investigator, General Hospital Groeninge
Other Study IDs: AZGS2018106
Record Dates: First submitted 2019-02-25; First posted 2019-02-27 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Oncology; Haematological Malignancy
Keywords: PAC infections; oncology
MeSH Terms: conditions — Neoplasms; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Removal of a central venous access device — We are interested in those patients for which a central venous access device was removed.

SUMMARY:
Background:

Central venous catheters are frequently used during cancer treatment with the aim of venepreservation. It can facilitate venous access for the safe administration of irritating or vesicant intravenous cancer medications and / or other fluids, to collect blood samples or to ensure accurate venous access for contrast during medical imaging. In addition, this means more comfort for the patient who needs to be punctured less peripherally. However, central venous catheters can also be a source of bloodstream infections and other complications, leading to increased morbidity and hospital costs (1). In our hospital, there is a general practice that if an infection of the device is suspected, the central venous catheter should be removed if antibiotics do not seem or prove to be effective.

The objective of this trial is to assess the frequency of implanted port catheter-removal in cancer patients due to suspected infection of the device in a particular oncology center over a time period of seven years. Furthermore, evidence for real device infections (per/post-surgery) and the potential contribution of different (institution-specific) risk factors on device infection will be explored. There will be focused on implanted port catheters only, as this is the main used central venous access device within the oncological population.

Trial objectives:

The primary aim of this retrospective descriptive trial is to evaluate the frequency of implanted port catheter-removal in cancer patients due to suspected infection of the device, over a time period of seven years.

The secondary aim is to examine whether the device infection could be confirmed during or after removal of the device.

At last, the tertiary aim is to verify whether certain variables can be denoted as potential risk factors for central venous access infection. Selection of those variables of interest will be based on a thorough review of the literature and discussion with the responsible healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

* Central venous access device removal in our general hospital
* Cancer patient

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We are interested in cancer patients who were implanted a central venous access device with regard to their cancer treatment, but for which the device was removed.
Sampling Method: Probability Sample
Enrollment: 1402 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Suspected infection rate | 2012-2017
  How many central venous access devices are removed due to a suspected infection of the device in cancer patients.

SECONDARY OUTCOMES:
Approved infection rate | 2012-2017
  For how many of the central venous access devices that were removed due to suspected infection of the device could an infection be confirmed?
Risk factors for central venous access device infections in cancer patients | 2012-2017
  Is it possible to denote certain variables as potential risk factors for central venous access device infection?

CONTACTS AND LOCATIONS:
Locations (1):
- GHGroeninge, Kortrijk, Belgium

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made publically and shared with other researchers.